CLINICAL TRIAL: NCT03466177
Title: Multimodal Retinal Imaging in the Detection and Follow-up of Alzheimer's Disease
Acronym: RetAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S60932
Record Dates: First submitted 2018-01-22; First posted 2018-03-15 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Alzheimer Disease; Alzheimer Dementia; Mild Cognitive Impairment; Dementia; Glaucoma; Age-Related Macular Degeneration; Diabetic Retinopathy
Keywords: Alzheimer's disease; Dementia; Mild cognitive impairment; Optical coherence tomography; Hyperspectral imaging; Multimodal retinal imaging
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia; Glaucoma; Macular Degeneration; Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Ab+ AD patients: amyloid positive Alzheimer's Disease patients
  - Ocular examination Visual acuity, biomicroscopy, funduscopy Fundus pictures, including hyperspectral imaging OCT + angio-OCT (Non-invasive, multimodal retinal imaging), Dynamic Vessel Analyzer (DVA)
  Interventions: Diagnostic Test: Non-invasive, multimodal retinal imaging
- Ab+ Mild Cognitive Impairment (MCI) patients: amyloid positive Mild Cognitive Impairment patients
  - Ocular examination Visual acuity, biomicroscopy, funduscopy Fundus pictures, including hyperspectral imaging OCT + angio-OCT (Non-invasive, multimodal retinal imaging), Dynamic Vessel Analyzer (DVA)
  Interventions: Diagnostic Test: Non-invasive, multimodal retinal imaging
- Ab+ cognitively intact volunteers: amyloid positive cognitively intact volunteers
  - Ocular examination Visual acuity, biomicroscopy, funduscopy Fundus pictures, including hyperspectral imaging OCT + angio-OCT (Non-invasive, multimodal retinal imaging), Dynamic Vessel Analyzer (DVA)
  Interventions: Diagnostic Test: Non-invasive, multimodal retinal imaging
- Ab- cognitively intact volunteers: amyloid negative cognitively intact volunteers
  - Ocular examination Visual acuity, biomicroscopy, funduscopy Fundus pictures, including hyperspectral imaging OCT + angio-OCT (Non-invasive, multimodal retinal imaging), Dynamic Vessel Analyzer (DVA)
  Interventions: Diagnostic Test: Non-invasive, multimodal retinal imaging
- Glaucoma patients: - Ocular examination Visual acuity, biomicroscopy, funduscopy Fundus pictures, including hyperspectral imaging OCT + angio-OCT (Non-invasive, multimodal retinal imaging), Dynamic Vessel Analyzer (DVA)
  Interventions: Diagnostic Test: Non-invasive, multimodal retinal imaging
- Age-related macular degeneration patients: - Ocular examination Visual acuity, biomicroscopy, funduscopy Fundus pictures, including hyperspectral imaging OCT + angio-OCT (Non-invasive, multimodal retinal imaging), Dynamic Vessel Analyzer (DVA)
  Interventions: Diagnostic Test: Non-invasive, multimodal retinal imaging
- Diabetic retinopathy patients: - Ocular examination Visual acuity, biomicroscopy, funduscopy Fundus pictures, including hyperspectral imaging OCT + angio-OCT (Non-invasive, multimodal retinal imaging), DVA
  Interventions: Diagnostic Test: Non-invasive, multimodal retinal imaging

INTERVENTIONS:
Diagnostic Test: Non-invasive, multimodal retinal imaging — Ocular exam including the application of different non-invasive ocular imaging techniques

SUMMARY:
Because of a shared ontogenic origin, the retina displays similarities to the brain and spinal cord in terms of anatomy, functionality, response to insult, and immunology. Hence, the retina can be approached as an integral part of the central nervous system. The occurence of ocular manifestations in several neurodegenerative pathologies, such as Alzheimer's disease and Parkinson's disease, accentuates the strong relationship between eye and brain. Particularly retinal changes can present a substrate for cerebral changes in these disorders. Offering a 'window to the brain', the transparent eye enables non-invasive imaging of these changes in retinal structure and vasculature. In this project, the potential of retinal biomarkers for e.g. Alzheimer's will be explored with the aim to overcome some of the hurdles in the current management of these pathologies, mainly the lack of techniques for patient screening and early diagnosis. The aim of this clinical trial is to correlate the retinal biomarkers for Alzheimer's with neuro-imaging, and cognitive function. Integrating the results will yield non-invasive retinal biomarkers for clinical research, screening, and follow-up of disease progression in various neurodegenerative disorders.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is the most common neurodegenerative disorder and the leading cause of dementia worldwide. A growing number of people are surviving into their 80s-90s and the number of AD patients projected to nearly triple in the next three decades, affecting 80-90 million people worldwide by 2040. As such, AD will become the third cause of death for older people, just behind cardiovascular disease and cancer. In contrast to the latter, AD cannot be prevented, slowed or cured. AD represents an enormous socio-economic burden and has become a trillion dollar disease. Despite decades of intensive research, diagnosis and treatment remain challenging for AD. A string of recent failures in clinical trials for AD drugs has pointed out that our understanding of the disease is still far from complete. More in detail, three major reasons underlying this treatment gap have been identified:

i. The lack of techniques for patient screening and early diagnosis. ii. The incomplete understanding of the complex interplay of pathological processes that underlie AD.

iii. The many hurdles between drug discovery and approval.

With this study, the investigators propose a novel way to address these needs, by using the retina as a model organ to study the central nervous system (CNS). Many of the hallmark cerebral pathophysiological processes of AD have also been observed in the retina. Unlike the rest of the CNS, the retina can be visualized directly, with an imaging resolution up to 100x higher than PET and MRI scans. Using these high-resolution imaging tools such as Optical Coherence Tomography (OCT), studies have demonstrated microvascular changes and neuro-retinal thinning in AD patients. Pilot data show that retinal Aβ can be visualized non-invasively solely based on the intrinsic hyperspectral signature of aggregated amyloid deposits. Non-invasive retinal imaging (e.g., fundus photography, OCT, hyperspectral imaging (HSI)) - which are all available at affordable cost -, could therefore represent novel means for identifying patients at risk, for longitudinal follow-up of disease progression in AD patients, and for research in a quest for more effective treatments.

This is an open-label longitudinal biomarker study without investigational medicinal product in subjects in different stages of the AD spectrum.

The data that we will collect consist of amyloid imaging, MRI, blood, genetic, general health and cognitive data, as well as visual acuity, ocular biomicroscopy and funduscopy, fundus photographs, hyperspectral retinal images, Optical Coherence Tomography (OCT) retinal images and OCT angiography (OCT-A) retinal images. Subjects will be followed longitudinally. In the current study the investigators will primarily investigate the potential of non-invasive, multimodal retinal imaging for the early detection of Alzheimer's disease and for the evaluation of disease progression. This will be done in comparison with amyloid imaging and neuropsychological evaluations.

The investigators will build a longitudinal database of ocular, systemic, neuro-psychiatric, MRI and PET imaging parameters of Aβ-positive and Aβ-negative patients with different stages of cognitive impairment. This database will be used to provide proof-of-concept that retinal biomarkers provide an early, accurate and non-invasive tool for AD detection and follow-up. All data will be collected in a database for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Between ≥ 50 and ≤ 85 years of age.
* In the opinion of the investigator, the patient is in stable medical condition and willing and able to perform study procedures.
* Patient is fluent in written and verbal Dutch.
* Patient is capable of giving informed consent.

Exclusion Criteria:

* Patient has a history or current evidence of a neurological disorder, which, in the opinion of the primary investigator, may contribute to the subject's cognitive impairment.
* Patient has a history of large-vessel stroke or evidence of a large-vessel infarction or other focal lesions on baseline MRI scan, which may contribute to the cause of the memory impairment in the opinion of the investigator. Vascular white matter lesions or other signs of microangiopathy will not be considered an exclusion.
* Patient has a history of malignancy ≤ 5 years prior to signing informed consent, except for patients who have undergone potentially curative therapy with no evidence of recurrence for 1 year, and who are deemed at low risk for recurrency by her/his treating physician.
* Patient is currently participating or has participated in a study with an investigational compound within 30 days of signing informed consent.
* Subject has any magnetizable metal prostheses, implants or foreign objects that could pose a hazard during MRI scans.
* Patient has a known history of ocular diseases other than the exception of cataract and/or wearing glasses/contact lenses.

Ages: 50 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Cfr. eligibility criteria
Sampling Method: Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Retinal biomarkers for AD: specificity | 5 years
  To evaluate the diagnostic performance of selected ocular biomarkers for Alzheimer's disease
Retinal biomarkers for AD: sensitivity | 5 years
  To evaluate the diagnostic performance of selected ocular biomarkers for Alzheimer's disease
Retinal biomarkers for AD: number needed to image | 5 years
  To evaluate the diagnostic performance of selected ocular biomarkers for Alzheimer's disease
Retinal biomarkers for AD: area under the curve (AUC) | 5 years
  To evaluate the diagnostic performance of selected ocular biomarkers for Alzheimer's disease
Retinal biomarkers for AD: receiver operating characteristic (ROC) | 5 years
  To evaluate the diagnostic performance of selected ocular biomarkers for Alzheimer's disease

SECONDARY OUTCOMES:
Retinal biomarkers for AD: quantification of cerebral Aβ load by non-invasive retinal imaging against the cerebral Aβ load measured by cerebral imaging | 15 years
  To deliver a proof-of-concept for the use of retinal biomarkers to quantitatively measure cerebral Aβ load by comparing the results of cerebral imaging (Standard Uptake Value ratio (SUVr) on amyloid-PET) with the results of retinal hyperspectral imaging (area of retinal Aβ detected, in µm²)
Retinal biomarkers for AD: disease progression by measuring the change from baseline at 2 years and more | 15 years
  To deliver a proof-of-concept for the use of retinal biomarkers to follow Alzheimer's disease progression by measuring the change from baseline at 2 years and after and to compare the results of the cerebral imaging and neuropsychiatric tests with the results from the selected retinal biomarkers for AD at different time points (t0, t 6 months, t 12 months, t 18 months, t 24 months, yearly for 15y)

CONTACTS AND LOCATIONS:
Overall Officials: Ingeborg Stalmans, MD PhD, Principal Investigator — UZ Leuven/KU Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2017-10-27): https://cdn.clinicaltrials.gov/large-docs/77/NCT03466177/Prot_000.pdf